

# SAP LYMA101 (PHASE II STUDY)

# LyMa101

Phase II study to evaluate the efficacy of upfront obinutuzumab in mantle cell lymphoma patients treated by DHAP followed by autologous transplantation plus obinutuzumab maintenance then MRD driven maintenance

# **Statistical Analysis Plan**

LYSARC: The Lymphoma Academic Research Organisation

⊠: Centre Hospitalier Lyon Sud – Bâtiment 2D

69495 Pierre Bénite Cedex - France

Version 2.0, the 09th of October 2024

| COORDINATING INVESTIGATOR | Pr Steven LE GOUILL |
|------------------------------|---------------------|
| CO-COORDINATING INVESTIGATOR | Pr Olivier HERMINE |
| COORDINATION CENTER | LYSARC |

| Initial Version and date of Protocol | Version 1.0 – May 09 <sup>th</sup> , 2016 |
|---|---|
| Last version and date of Protocol | Version 5.0 – April 04 <sup>th</sup> , 2018 |
| EudraCT Number | 2016-000548-33 |

| BIOSTATISTICS | Samuel GRIOLET<br>LYSARC |
|---|---|
| | CHU Lyon Sud Bât. 2D<br>69495 Pierre-Bénite - France<br>samuel.griolet.ext@lysarc.org |

# **APPROVAL PAGE**

| | Signature | Date |
|---|---|---|
| Pr LE GOUILL Steven, Coordinating Investigator | | |
| Pr HERMINE Olivier, Co-coordinating Investigator | | |
| PLEAU-PISON Thomas, Clinical Project Manager | | |
| <b>BENKHALFALLAH Asma</b> , Biology project manager | | - |
| GRIOLET Samuel LYSARC Biostatistician | grobe | 05 DFC 2024 |

# **Document History:**

| Version # | Effective Date | Author | Modification Description | Affected |
|---|---|---|---|---|
| | | | | Paragraphs |
| 1.0 | 11JAN2019 | Samuel GRIOLET | | |
| 2.0 | 09OCT2024 | Samuel GRIOLET | Maintenance on demand added Analysis of MRD during maintenance | |

# **TABLE OF CONTENTS**

| Li | st of A | bbre | viations | 6 |
|---|---|---|---|---|
| 1 | Intr | oduc | tion | 7 |
| 2 | Inve | estiga | ational plan | 8 |
| | 2.1 | Ratio | onale | . 8 |
| | 2.2 | Stud | ly Design | . 9 |
| 3 | Stud | dy ok | pjectives and endpoints 1 | ΙΟ |
| | 3.1 | Obje | ectives | 10 |
| | 3.1.1 | L | Primary objective | 10 |
| | 3.1.2 | 2 | Secondary objectives | 10 |
| | 3.1.3 | 3 | Exploratory objectives | 10 |
| | 3.2 | Eval | uation endpoints | 10 |
| | 3.2.1 | L | Primary efficacy endpoint | 10 |
| | 3.2.2 | | Secondary efficacy endpoints | |
| | 3.2.3 | | Secondary safety endpoints | |
| | 3.2.4 | ŀ | Exploratory endpoints | 12 |
| | 3.3 | Follo | ow-up duration | 13 |
| | 3.4 | Exte | nt of exposure | 13 |
| 4 | Stat | istic | al Considerations 1 | L <b>4</b> |
| | 4.1 | Sam | ple size calculation | 14 |
| | 4.2 | Prim | nary criterion analysis | 14 |
| | 4.3 | Fina | l analysis | 15 |
| | 4.4 | Anal | lysis Sets | 15 |
| | 4.4.1 | L | Included Set (IS) | 15 |
| | 4.4.2 | <u>)</u> | Efficacy Set (ES) | |
| | 4.4.3 | | Modified Efficacy Set (mES) | |
| | 4.4.4 | ļ | Safety Set (SS) | 15 |
| | 4.5 | Gen | eral statistical approach | 15 |
| | 4.5.1 | L | Statistical analysis | 15 |
| | 4.5.2 | <u>)</u> | Statistical methods | |
| | 4.5.3 | 3 | Statistical Approach for control of Alpha | 16 |
| | 4.6 | Han | dling of missing or off-schedule data | 16 |
| | 4.7 | Soft | ware | 16 |
| 5 | Stat | istic | al outputs 1 | L <b>7</b> |
| | 5.1 | Stud | ly summary | 17 |
| | 5.1.1 | | Overall description | |
| | 5.1.2 | | Study dates | |
| | 5.1.3 | _ | Follow-up duration | |
| | 5.2 | Stud | ly patients | 10 |
| | 5.2.1 | | Disposition of patients | |
| | 5.2.2 | - | Analysis sets | |
| | | - | usion / Exclusion criteria | |
| | 3.5 | INCIL | JS1011 / EXCIUSION CITLENA | ۷3 |

| | 5.4 | Protocol deviations | 24 |
|---|---|---|---|
| | 5.5 | Demographic and other baseline characteristics | 24 |
| | 5.5.1 | | |
| | 5.5.2 | Nodal involvement | 25 |
| | 5.5.3 | B Extra-nodal involvement | 27 |
| | 5.5.4 | 4 Bone Marrow | 29 |
| | 5.5.5 | 5 Staging | 29 |
| | 5.5.6 | 6 MRD | 29 |
| | 5.6 | Evaluation during study | 30 |
| | 5.6.1 | • | |
| | 5.6.2 | | |
| | 5.6.3 | | |
| | 5.7 | Efficacy Analysis | 31 |
| | 5.7.1 | | |
| | 5.7.2 | | |
| | 5.7.2 | | |
| | 5.7.4 | | |
| | 5.7.5 | | |
| | 5.7.6 | | |
| | 5.7.7 | | |
| | 5.7.8 | · · | |
| | 5.8 | Progression / Relapse | |
| | 5.9 | Extent of exposure | 38 |
| | 5.9.1 | | |
| | 5.9.2 | 2 Dose | 39 |
| | 5.10 | Safety analysis | 42 |
| | 5.10. | • | |
| | 5.10. | .2 Serious Adverse Events | 44 |
| | 5.10. | | |
| | 5.10. | | |
| | 5.10. | | |
| | - 44 | · | |
| | 5.11 | | |
| | | .1 Concomitant treatments at inclusion | |
| | 5.11. | .2 Concomitant treatments during treatment period | 51 |
| | 5.12 | Non study treatments out of progression | 51 |
| 6 | Refe | erences | 53 |
| 7 | <b>∆</b> ppr | ENDICES | E/I |
| , | | | |
| | 7.1 | Demographic and other baseline characteristics | 54 |
| | 7.2 | Evaluation during study | <b>56</b> |
| | 7.3 | Appendix A: Calculation of total dose and PPD | <b>56</b> |
| | 7.4 | Appendix B: MCL International Prognostic Index (MIPI) and combined biological Index | |
| | | )) | <b>57</b> |
| | ·<br>7.5 | Appendix C: Response Criteria for Lymphoma – Lugano Classification | |
| | | LL | |

### LIST OF ABBREVIATIONS

AE Adverse Event

AEPI Adverse Event of Particular Interest
AESI Adverse Event of Specific Interest
ASCT Autologous Stem Cell Transplant

BM Bone Marrow
BSA Body Surface Area

CHOP Cyclophosphamide, doxorubicin, vincristine, and prednisone

CI Confidence Interval
CR Complete Response
CRR Complete Response Rate

CRu Complete Response unconfirmed

CT Computed Tomography

CTCAE Common Terminology Criteria for Adverse Events

DOR Duration Of Response

ECOG Eastern Cooperative Oncology Group

EFS Event-Free Survival

FLIPI Follicular Lymphoma International Prognostic Index

G-CSF Granulocyte Colony-Stimulating Factor

HBV Hepatitis B virus HCV Hepatitis C virus

HIV Human immunodeficiency virus

ICF Informed Consent Form

IDMC Independent Data Monitoring Committee

IRR Infusion Related Reaction
LDH Lactic DeHydrogenase
MCL Mantle Cell Lymphoma
MRD Minimal Residual Disease
NCI National Cancer Institute

ND Not Done

NHL Non-Hodgkin's Lymphoma
ORR Overall response Rate
OS Overall Survival
PD Progressive Disease

PET <sup>18</sup>F-FDG Positron Emission Tomography

PFS Progression Free Survival
PI Principal Investigator

PPD Percentage of Planned Dose

PR Partial Response
PS Performance Status
PT Preferred Term
QoL Quality Of Life

SAE Serious Adverse Event SAP Statistical Analysis Plan

SD Stable Disease
SOC System Organ Class
OPM Other Primary Malignancy

LYSARC 

# 1 Introduction

This document describes the statistical analyses and the different layouts for tables and listings to be produced for the protocol **LyMa101** titled "Phase II study to evaluate the efficacy of upfront obinutuzumab in mantle cell lymphoma patients treated by DHAP followed by autologous transplantation plus obinutuzumab maintenance then MRD driven maintenance".

One interim analyse for the primary criterion is planned for this study.

The statistical analysis plan (SAP) provides a comprehensive and detailed description of the strategy, rationale, and statistical methods to be applied to assess the efficacy and safety of Obinutuzumab (GA101), in patients with previously untreated MCL treated by DHAP.

The purpose of the SAP is to ensure the credibility of the study findings by pre-specifying the statistical approaches for all data analysis before database lock.

The SAP is finalized and signed prior to the clinical database lock.

LYSARC 

# 2 INVESTIGATIONAL PLAN

#### 2.1 Rationale

Achievement and preservation of minimal residual disease (MRD) response is the strongest independent predictor of prognosis in MCL patients. By using MRD status as tool for treatment selection, treatment should be focused to achieve and maintain a maximum MRD response to improve outcome. (Pott Blood 2010, Abstract ASH 2014).

Because of the economic constraints of maintenance therapy, preemptive treatment using rituximab based on MRD relapse should be evaluated and might be effective at preventing clinical relapse. Indeed, it has been shown in 32 MCL patients that MRD-based preemptive rituximab therapy restored a PCR-negative state in 81% of cases, of whom 38% subsequently relapsed clinically at a median time of 3.9 years (Andersen JCO 2009, Geisler BJH 2012). Pre-emptive treatment may thus prevent relapse in at least some patients and may prove to be a more cost effective strategy. Use of pre-emptive treatment requires definition of molecular relapse, which is classically based on a progressive rise in MRD levels in three consecutive samples, which can be increasingly closely spaced.

The gold standard for monitoring MRD in MCL is real-time quantitative polymerase chain reaction (RQ-PCR) amplification of clonal immunoglobulin heavy chain (IgH) VDJ or IgH-BCL1 rearrangements, which are informative in 90% and 40% of patients respectively (Pott Blood 2006, Andersen JCO 2009). RQ-PCR strategies are sufficiently sensitive (minimum 0.01%) and specific for MRD quantification in around 85% of MCL patients. These strategies are, however, long, complex and associated with a significant grey zone of non-quantifiable positivity, Below the Quantitative Range (BQR). The quantifiable range (QR) should ideally be at least 0.01% (10E-4), but this is not achieved in 20-25% of samples (Cheminant et al. submitted). For these reasons, RQ-PCR is increasingly challenged by multicolor Flow cytometry (MFC) or droplet digital PCR (ddPCR).

Approximately 10% of MCL patients are not accessible to RQ-PCR MRD with acceptable sensitivity and QR. A proportion of these cases become accessible to MRD assessment by MFC (Cheminant, submitted) or by PCR quantification relative to patient specific plasmid calibrators (Gimenez et al. BJH 2012). The use of MRD results for patient stratification obviously requires maximal informativity. Therefore, the present project will also investigate complementary techniques, including MFC, ddPCR and/or plasmid calibrators.

During follow-up, the percentage of MRD positive samples was approximately 20-25% during the first 3 years, and less than 20% at later time points (Pott ASH 2014 abstract 147). Among patients with clinical relapses, it has been shown that clinical relapse is strongly associated with MRD positivity. In an analysis of the EU-MCL network, only 13% of MCL patients were peripheral blood (PB)-negative (Pott ASH 2014 abstract 147), whereas this will be the predominant source of material for MRD analysis in the proposed study, for ease of sampling, patient comfort and because informativity is comparable to bone marrow analysis, particularly at later time points.

To the present trial will determine what proportion of patients' clinical relapse is preceded by molecular relapse and with what delay. In the EU-MCL studies, the latency between the first positive MRD and the clinical relapse varies greatly between patients. The median latency for prediction by RQ-PCR when any increase to at least 2 positive triplicates was considered as MRD relapse was 22.5 months [range 1-48m] and 5 months [range 2-11m] when only results above 0.01% were considered positive, with no difference between RQ-PCR and MFC quantification (Cheminant et al. submitted).

LYSARC 

# 2.2 Study Design



LYSARC 

# **3** STUDY OBJECTIVES AND ENDPOINTS

# 3.1 Objectives

#### 3.1.1 Primary objective

The primary objective of the study is to evaluate the efficacy of upfront Obinutuzumab (GA101) at the molecular level (MRD) in bone marrow after induction, after the 4 cycles or at premature discontinuation, in patients with previously untreated MCL treated by DHAP..

#### 3.1.2 Secondary objectives

The secondary objectives of the study are:

- To evaluate the efficacy of the obinutuzumab in patients with MCL treated by DHAP before ASCT, after ASCT and every 6 months in terms of clinical response (Cheson 99) and MRD plus in terms of FDG-PET before and after ASCT
- To evaluate PFS, Overall survival at study end
- To evaluate the incidence of stem cell collection failure after obinutuzumab-DHAP = GA-DHAP
- To evaluate MRD negativity after 3 years of maintenance and maintenance "on-demand"
- To evaluate PET results after 3 years of maintenance
- Duration of MRD negativity
- To evaluate tolerability of obinutuzumab at induction and then "on-demand"

### 3.1.3 Exploratory objectives

The exploratory objectives of the study is:

• To determine baseline prognostic factors on PFS and OS

# 3.2 Evaluation endpoints

#### 3.2.1 Primary efficacy endpoint

The primary endpoint is the Molecular residual disease (MRD) negativity after induction. Assessment of MRD will be based on molecular level in BM according to EU MCL network guidelines. Patient without MRD assessment (due to whatever reason) will be considered as MRD positive. This endpoint will be analyzed on efficacy set (ES) and also on modified efficacy set (mES) as sensitivity analysis.

LYSARC 

#### 3.2.2 Secondary efficacy endpoints

The following secondary efficacy endpoints will be analyzed using appropriate statistical methods.

#### 3.2.2.1 Secondary efficacy endpoint 1

#### Response according to Cheson 99 and overall response rate after 3 years of maintenance

Response after 3 years of maintenance will be evaluated. Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 1999)). Patient without response assessment (due to whatever reason) will be considered as non-responder. Overall (CR/PR) response rate will be also presented.

An additional analysis will be performed considering as non-responders all patients who relapsed or died during treatment phase even if they were prematurely treatment discontinued as responder during treatment phase.

This endpoint will be analyzed on efficacy set (ES) and on safety set (SS).

#### 3.2.2.2 Secondary efficacy endpoint 2

#### PET result after 3 years of maintenance

PET result after 3 years of maintenance will be evaluated. Assessment of PET will be based on Lugano 2014 criteria (according to Cheson & Al. J. Clinic Oncol 2015). See Appendix C (Reponse criteria for lymphoma – Lugano classification).

This endpoint will be analyzed on efficacy set (ES) and on safety set (SS).

#### 3.2.2.3 Secondary efficacy endpoint 3

# MRD after 3 years of maintenance and after maintenance "on demand"

Molecular residual disease (MRD) after 3 years of maintenance and after maintenance "on demand" will be evaluated. Assessment of MRD will be based on molecular level in BM according to EU MCL network guidelines. Patient without MRD assessment (due to whatever reason) will be considered as MRD positive.

This endpoint will be analyzed on efficacy set (ES).

#### 3.2.2.4 Secondary efficacy endpoint 4

#### **PFS**

PFS is defined as the time from inclusion into the study to the first observation of documented disease progression or death due to any cause. If a subject has not progressed or died, PFS will be censored at the time of last visit with adequate assessment.

This endpoint will be analyzed on efficacy set (ES) and on safety set (SS).

## 3.2.2.5 Secondary efficacy endpoint 5

#### OS

Overall survival will be measured from the date of inclusion to the date of death from any cause. Alive patients will be censored at their last contact date.

This endpoint will be analyzed on efficacy set (ES) and on safety set (SS).

LYSARC 

#### 3.2.2.6 Secondary efficacy endpoint 6

#### Stem cell collection failure

Stem cell collection failure will be evaluated after induction.

This endpoint will be analyzed on efficacy set (ES) and on safety set (SS).

#### 3.2.2.7 Secondary efficacy endpoint 7

# **Duration of MRD negativity**

Duration of MRD negativity is defined as the time from the date of attainment the first negative MRD to the date of positive MRD. Duration or MRD negativity would be assessed for patients with at least one MRD negativity and as survival endpoint. For patients achieving a negative MRD but who have not positive MRD or not MRD assessment at the time of analysis, duration of MRD negativity will be censored on the date of last MRD assessment.

This endpoint will be analyzed on efficacy set (ES).

#### 3.2.3 Secondary safety endpoints

Summary of study drug administration including treatment duration and average dose will be displayed.

Number, frequency, reasons for premature treatment discontinuation and study discontinuation will be summarized.

Adverse events, clinical laboratory measurements will be described.

AEs will be classified using the latest version of Medical Dictionary for Drug Regulatory Activities (MedDRA) coding system at the time of database lock. The severity of the toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) whenever possible. Subsets of AEs to be summarized include serious, NCI CTCAE grade severities, suspected treatment-related, and events that resulted in withdrawal of investigational product. The most severe grade of each preferred term for a patient will be utilized for summaries of adverse events by NCI CTCAE grade.

All AEs and SAEs will be described by system organ class and preferred term (a patient having the same event more than once will be counted only once) by period. Focus on AEs leading to death, Aes leading to discontinuation from treatment and AEs of special interest (i.e Tumor Lysis Syndrom) will also be displayed in a separate table and listing.

All deaths will be listed and summarized by cause of death and narratives of death will be also presented.

This endpoint will be performed on safety set (SS).

#### 3.2.4 Exploratory endpoints

The following exploratory endpoint will be summarized using appropriate statistical methods.

#### **Baseline prognostic factors on PFS and OS**

A dedicated analysis on survival (PFS/OS) will be performed in order to determined baseline prognostic factors. The implemented method will take into account the specificities of on-demand treatment during the second maintenance period.

LYSARC 

# 3.3 Follow-up duration

The follow-up duration is defined as the time between the inclusion date and the last contact date. Follow-up duration is based on OS and calculated with a reverse Kaplan-Meier method. Deceased patients are censored at the date of death.

# 3.4 Extent of exposure

- Treatment duration
- Total dose
- % planned dose

LYSARC 

# 4 STATISTICAL CONSIDERATIONS

# 4.1 Sample size calculation

#### **Hypothesis:**

We expect to have an increase of 15% of the MRD negativity in bone marrow (BM) rate for patients treated with GA-DHAP.

Based on the interim results of LYMA presented at ASH 2014, the MRD negativity rate were 65% (Legouill, ASH 2014). Nevertheless, in the LYMA study, the MRD has been assessed after 4 cycles of DHAP only for patient that completed the 4 cycles. Therefore this rate does not take into account the rate of patients who progressed on treatment or took R-CHOP because of insufficient response. If we take into account these patients considering them as non responder patients and based on the LYSA/LYSARC experience, then the MRD negativity rate of all patients in the LYMA may be around 55%. Considering that these patients will also be included in the LyMa101 we have to take into account a rate of 55% of MRD negativity instead of 65% in the sample size calculation.

The hypotheses are as follows:

- Experimental treatment will be considered ineffective if the MRD negativity in BM after the 4 cycles or at treatment discontinuation (at a molecular level) proportion is ≤ 55% (P<sub>0</sub>)
- Experimental treatment will be considered effective if the MRD negativity in BM after the 4 cycles or at treatment discontinuation (at a molecular level) proportion ≥ 70% (P₁)
- $\alpha$  risk of 0.05 and  $\beta$  of 0.20
- one-sided test

Patients will be considered as MRD positive if the patient has no MRD assessment due to whatever the reason.

#### Sample Size:

A total of 70 evaluable patients will be required for this study. Assuming that some included patients will not receive the treatment or will not be informative for MRD in bone marrow and/or blood at baseline, enrollement will be done until 70 patients are evaluable. For this purpose, about 83 patients should be enrolling (15% drop-out).

Sample size calculation was performed using an exact single-stage phase II design with East 5.4 (A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med. 2001. 20(6):859-66).

# 4.2 Primary criterion analysis

This analysis will be performed once all patients included in efficacy set (70 patients) have completed the 4 cycles of treatment or treatment discontinued prior to cycle 4 and will consist of analyzing:

- Primary criterion: MRD negativity in BM rate after the 4 cycles or at treatment discontinuation of GA-DHAP
- Treatment exposure
- Stem cell collection failure
- Secondary safety endpoints

LYSARC 

Among the 70 evaluable patients, if 46 patients or more have a MRD negativity after the 4 cycles or at treatment discontinuation the treatment will be considered as sufficiently effective and further investigations (another trial) will have to be foreseen.

# 4.3 Final analysis

This analysis will be performed when all included patients will undergo the end of treatment visit (at end of maintenance "on demand" period or at treatment discontinuation) and will consist of the whole statistical analyses.

At this time all secondary and exploratory endpoints will be analyzed.

### 4.4 Analysis Sets

#### 4.4.1 Included Set (IS)

The included set will include all included patients having signed the informed consent.

#### 4.4.2 Efficacy Set (ES)

The Efficacy set will include all patients having signed the informed consent, received at least one dose of the IMP study drug (Obinutuzumab) and with an informative MRD in BM and/or blood at baseline.

#### 4.4.3 Modified Efficacy Set (mES)

The modified Efficacy Set will include all patients having signed the informed consent, received at least one dose of the IMP study drug (Obinutuzumab), with an informative MRD in BM and/or blood at baseline and an informative MRD in BM after the 4 cycles of GA-DHAP or at treatment discontinuation.

#### 4.4.4 Safety Set (SS)

The Safety set will include all patients having signed the informed consent and received at least one dose of the IMP study drug (Obinutuzumab).

#### 4.5 General statistical approach

## 4.5.1 Statistical analysis

<u>Continuous data</u> will be summarized in tables displaying number of observations, mean, standard deviation, median, range; quartiles will also be presented when considered relevant.

<u>Categorical data</u> will be expressed as frequencies and percentages (of non-missing data).

Response rates (according to Cheson 1999 or MRD) will be expressed with 90% confidence limits (to be consistent with one sided 5% level of significance) according to Pearson-Clopper method. The number and percent of patients falling into each category of response will be provided.

<u>Time to event</u> will be performed using Kaplan-Meier method. Survival probabilities, median survival and quartiles will be estimated with their 95% CI. Survival curves will be provided. A dedicated analysis on survival (PFS/OS) will be performed in order to determined baseline prognostic factors. The implemented method will take into account the specificities of on-demand treatment during the second maintenance period.

LYSARC 

#### 4.5.2 Statistical methods

Unless otherwise noted, statistical tests will be two-sided and performed using a 5% level of significance.

The Kaplan Meier method<sup>1,3</sup>, also known as the "product-limit method", is a non-paramatric method for estimating the probability of survival at any given point in time. The kaplan-meier method handles both censored and uncensored data.

The log-rank test<sup>1</sup> is a non-parametric test for comparing the survival distributions of two or more groups. This test is computed using the expected and observed number of events in each group.

Cox proportional-hazard model<sup>1,2,3</sup> is a semi-parametric model used for testing differences in survival times of two or more groups of interest, while allowing to adjust for covariates of interest.

Chi-square test<sup>1</sup> is used to test equality of proportions between two or more populations and is computed by comparing the observed and expected counts when the null hypothesis is true.

The Wilcoxon rank-sum test<sup>1</sup>, also called Mann–Whitney U test, is a non-parametric test used to compare disrtibutions from two independent groups and assess whether one has systematically larger values than the other.

The independent samples T-Test<sup>3</sup> is a parametric test used to compare the means of a normally distributed variable for two independent groups.

Logistic regression<sup>1,3</sup> is a regression model in which the outcome is a categorical variable. The log odds of the outcome are modeled as a linear combination of the predictor variables.

#### 4.5.3 Statistical Approach for control of Alpha

No adjustment for multiple comparisons will be made.

#### 4.6 Handling of missing or off-schedule data

No imputation of values for missing data will be performed.

#### 4.7 Software

All outputs will be produced using SAS version 9.4 or higher and AdClin version 3.5.0 or higher.

LYSARC 

# **5** STATISTICAL OUTPUTS

# **5.1** Study summary

# 5.1.1 Overall description

Table 4.7-1 Global recruitment status

| | All patients |
|--------------|--------------|
| | N=XX |
| Included Set | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Table 4.7-2 Number of patients by center – Included Set

| | Included Set |
|-------------|--------------|
| | N=XX |
| Center Name | |
| Center X | XX (XX.X%) |
| Center X | XX (XX.X%) |
| | XX (XX.X%) |

Table 4.7-3 Number of patients at each timepoint – Included Set

| | Included Set |
|-----------------------------------------|--------------|
| | N=XX |
| Baseline | |
| Evaluation at baseline | XX (XX.X%) |
| Induction | |
| Cycle 1 | XX (XX.X%) |
| Cycle 2 | XX (XX.X%) |
| Cycle 3 | XX (XX.X%) |
| Cycle 4 | XX (XX.X%) |
| Evaluation after induction | XX (XX.X%) |
| ASCT | |
| ASCT | XX (XX.X%) |
| Evaluation after ASCT | XX (XX.X%) |
| Maintenance | |
| V1 | XX (XX.X%) |
| | XX (XX.X%) |
| V19 | XX (XX.X%) |
| Evaluation after 3 years of maintenance | XX (XX.X%) |
| Maintenance on-demand | |
| On-demand visit 1 | XX (XX.X%) |
| | XX (XX.X%) |
| On-demand visit 36 | XX (XX.X%) |
| End of treatment | |
| Evaluation at the end of treatment | XX (XX.X%) |

Table 4.7-4 Number of patients by follow-up interval – Included Set

| | Included Set |
|----------------------------|--------------|
| | N=XX |
| Follow-up visits performed | |
| FU n°1 | XX (XX.X%) |
| FU n°2 | XX (XX.X%) |
| | XX (XX.X%) |

LYSARC 

#### 5.1.2 Study dates

Table 4.7-1 Date of inclusion – Included Set

| | Included Set |
|-------------------------|--------------|
| | N=XX |
| Inclusion date | |
| Date of first inclusion | XX/XX/XXXX |
| Date of last inclusion | XX/XX/XXXX |

#### Table 4.7-2 Date of last visit\* last patient – Included Set

| | Included Set<br>N=XX |
|-------------------------------------|----------------------|
| Date of last visit* of last patient | XX/XX/XXXX |

<sup>\*</sup> Last visit includes visits performed during follow-up period

Table 5.1.2-3 Study duration\* – Included Set

| | Included Set |
|--------------------------|--------------|
| | N=XX |
| Study duration* (months) | |
| N | XX |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1 ; Q3 | XX ; XX |
| Min ; Max | XX ; XX |

<sup>\*</sup> Study duration is calculated from date of inclusion until date of last contact (including FU).

# 5.1.3 Follow-up duration

Figure 4.5.3-1 Follow up throughout the study<sup>(1)</sup> – Included set

Table 4.5.3-1 Follow up throughout the study<sup>(1)</sup> – Survival summary – Included set

| | N | Median | 95% CI lower | 95% CI Upper | Min | Max |
|---|---|---|---|---|---|---|
| Follow up duration (months) | XX | XX | XX | XX | XX | XX |

<sup>(1)</sup> Reverse Kaplan-Meier regression model on OS.

LYSARC 

<sup>(1)</sup> Reverse Kaplan-Meier regression model on OS

# 5.2 Study patients

#### **5.2.1** Disposition of patients

Figure 4.7-1 Disposition of patients



LYSARC 

Table 4.7-1 Premature treatment discontinuation – Included Set

| able 4.7-1 Premature treatment discontinuation – in | |
|---|---|
| | Included Set |
| | N=XX |
| Premature treatment discontinuation | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, reason | |
| Progressive Disease | XX (XX.X%) |
| Adverse Event | XX (XX.X%) |
| Death | XX (XX.X%) |
| Withdrawal by subject | XX (XX.X%) |
| Protocol deviation | XX (XX.X%) |
| Other | XX (XX.X%) |
| Lack of efficacy | XX (XX.X%) |
| Non-compliance with study drug | XX (XX.X%) |
| Physician decision | XX (XX.X%) |
| If yes, period | |
| Before treatment | XX (XX.X%) |
| Induction | XX (XX.X%) |
| ASCT | XX (XX.X%) |
| Maintenance | XX (XX.X%) |
| Follow-Up | XX (XX.X%) |
| If yes, time since inclusion (months) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

Listing 4.7-1 Premature treatment discontinuation – Included Set (XX patients)

| Patient identification | Date of | Premature treatment discontinuation | | | | |
|---|---|---|---|---|---|---|
| number | inclusion | Y/N | Date | Period | Reason | Description (eventually) |
| XXXXX | XX/XX/XXXX | XX | XX/XX/XXXX | XX | XXX | XXX |

Listing 4.7-2 Premature treatment discontinuation due to AEs – Included Set (XX patients)

| Patient identification | Date of | | Treatment | discontin | uation | Λ | dverse event |
|---|---|---|---|---|---|---|---|
| Patient identification | Date of | | пеашеш | uiscontiii | uation | A | uverse event |
| number | inclusion | Y/N | Date | Period | Reason | Description | Action taken on GA101 |
| XXXXX | XX/XX/XXXX | XX | XX/XX/XXXX | XX | Adverse Event | XX | XX |

Filter: Reason for treatment discontinuation = adverse event

LYSARC 

#### 5.2.2 Analysis sets

<u>The included set</u> will include all included patients having signed the informed consent.

<u>The Safety set</u> will include all patients having signed the informed consent and received at least one dose of the IMP study drug (Obinutuzumab).

<u>The Efficacy set</u> will include all patients having signed the informed consent, received at least one dose of the IMP study drug (Obinutuzumab) and with an informative MRD in BM and/or blood at baseline.

<u>The modified Efficacy Set</u> will include all patients having signed the informed consent, received at least one dose of the IMP study drug (Obinutuzumab), with an informative MRD in BM and/or blood at baseline and an informative MRD in BM after the 4 cycles of GA-DHAP or at treatment discontinuation.

Table 5.2.2-1 Analysis Sets – Included Set

| | Included Set |
|-----------------------|--------------|
| | N=XX |
| Safety Set | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Efficacy Set | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Modified Efficacy Set | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Listing 5.2.2-1 Patients excluded from Safety Set (XX patients)

| Patient identification | Safety Set | Inclusion date | Received at least | Number of cycles |
|---|---|---|---|---|
| number | | | one dose of GA101 | received |
| XXXXX | No | XX/XX/XXXX | XX | XX |

#### Listing 5.2.2-2 Patients excluded from Efficacy Set (XX patients)

| Patient<br>identification<br>number | Efficacy<br>Set | Inclusion<br>date | Received at least one cycle of GA-DHAP | Premature<br>withdrawal | MRD in BM at baseline | MRD in blood at baseline | Number of cycles received |
|---|---|---|---|---|---|---|---|
| XXXXX | No | XX/XX/XXXX | XX | XX | XX | XX | XX |

#### Listing 5.2.2-3 Patients excluded from Modified Efficacy Set (XX patients)

| Patient identification number | Modified<br>Efficacy Set | Inclusion<br>date | Received at least<br>one cycle of GA-<br>DHAP | Premature<br>withdrawal | MRD in BM at baseline | MRD in<br>blood at<br>baseline | MRD in<br>BM after 4<br>cycles | Number of cycles received |
|---|---|---|---|---|---|---|---|---|
| XXXXX | No | XX/XX/XXXX | XX | XX | XX | XX | XX | XX |

LYSARC 

Figure 5.2.2-1 Analysis Sets



LYSARC 

# 5.3 Inclusion / Exclusion criteria

Table 4.5.3-2 Patients with at least one criterion not fulfilled – Included Set

| | Included Set |
|--------------------------------------------------------------|--------------|
| | N=XX |
| Patients with at least one criterion not fulfilled | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Patients with at least one inclusion criterion not fulfilled | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Patients with at least one exclusion criterion not fulfilled | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Table 4.5.3-3 Inclusion Criteria – Included Set

| | Includ<br>N= | ed Set<br>XX |
|-----------------------|--------------|--------------|
| | Yes | No |
| Inclusion Criteria 1 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 2 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 3 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 4 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 5 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 6 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 7 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 8 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 9 | XX (XX.X%) | XX (XX.X%) |
| Inclusion Criteria 10 | XX (XX.X%) | XX (XX.X%) |

Table 4.5.3-4 Exclusion Criteria – Included Set

| | Included Set<br>N=XX | | |
|-----------------------|----------------------|------------|------------|
| | Yes | No | NA |
| Exclusion Criteria 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 5 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 6 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 7 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 8 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 9 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 10 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 11 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 12 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 13 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 14 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 15 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 16 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Exclusion Criteria 17 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Listing 4.5.3-1 Patients with inclusion and or exclusion criterion not fulfilled – Included Set (XX patients)

| Patient identification | Age | | Inclusion | Date of signature of consent | | Criterion not fulfilled | |
|---|---|---|---|---|---|---|---|
| number | (years) | Sex | date | | Number | Definition | Value of<br>criterion |
| XXXXX | XX | Х | XX/XX/XXXX | XX/XX/XXXX | XX | XX | Х |

LYSARC 

# **5.4 Protocol deviations**

Table 4.7-5 Major protocol deviations – Included Set

| | Included Set |
|---|---|
| | N=XX |
| Patients with at least one major protocol deviation | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, type of major protocol deviation | |
| Treatment received before the signature of informed consent | XX (XX.X%) |
| Non respect of inclusion criteria | XX (XX.X%) |
| Non respect of exclusion criteria | XX (XX.X%) |
| Diagnosis not validated with ANAPATH reviewed | XX (XX.X%) |
| No BM aspirate done for MRD analysis after induction or PWD | XX (XX.X%) |
| No BM aspirate done for MRD analysis after 3 year maintenance or PWD | XX (XX.X%) |
| MRD assessment not done during maintenance-on-demand | XX (XX.X%) |
| Positive MRD during maintenance-on-demand but no GA101 afterward | XX (XX.X%) |

# 5.5 Demographic and other baseline characteristics

Table 4.7-6 Summary of main baseline characteristics – Included Set

| | Included Set |
|----------------------------------------------|--------------|
| | N=XX |
| Sex | |
| Male | XX (XX.X) |
| Female | XX (XX.X) |
| Age at inclusion (years) | |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Ann Arbor stage | |
| II | XX (XX.X) |
| III | XX (XX.X) |
| IV | XX (XX.X) |
| Bio-MIPI | |
| Low risk | XX (XX.X%) |
| Intermediate risk | XX (XX.X%) |
| High risk | XX (XX.X%) |
| Performance status (ECOG) | |
| 0 | XX (XX.X) |
| 1 | XX (XX.X) |
| 2 | XX (XX.X) |
| 3 | XX (XX.X) |
| 4 | XX (XX.X) |
| Bulky Disease (cm) | |
| >= 5 | XX (XX.X) |
| < 5 | XX (XX.X) |
| Bone Marrow involvement (biospy or aspirate) | |
| Involved | XX (XX.X) |
| Not Involved | XX (XX.X) |
| Not Evaluable | XX (XX.X) |
| B symptoms | |
| No | XX (XX.X) |
| Yes | XX (XX.X) |
| Ki67 (%) | <u> </u> |
| >= 30% | XX (XX.X) |
| Median | xx.x |
| Min ; Max | XX;XX |
| Blastoid variant | |
| No | XX (XX.X) |
| Yes | xx (xx.x) |

LYSARC 

# 5.5.1 Diagnosis

Table 4.7.1-1 Diagnosis at baseline – Included Set

| | Included Set |
|-----------------------------------------------|--------------|
| | N=XX |
| Time between diagnosis and inclusion (months) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Pathological diagnosis | |
| Mantle Cell Lymphoma | XX (XX.X%) |
| Other histology non authorized | XX (XX.X%) |
| If Other, specify | |
| XXX | XX (XX.X%) |
| XXX | XX (XX.X%) |
| Pathological report | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Diagnosis (local) | |
| XXX | XX (XX.X%) |
| XXX | XX (XX.X%) |
| Diagnosis according to the central review | |
| XXX | XX (XX.X%) |
| XXX | XX (XX.X%) |
| Blastoid variant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Ki67 (%) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

#### 5.5.2 Nodal involvement

Table 4.7.2-1 Nodal involvement at baseline – Included Set

| 10010 11712 2 110001 111101101110111011011 | |
|----------------------------------------------|--------------|
| | Included Set |
| | N=XX |
| Patients with at least one nodal involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Table 4.7.2-2 Description of nodal involvement at baseline – Included Set

| | Included Set<br>N=XX |
|-----------------------|----------------------|
| Cervical Right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Cervical Left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Supraclavicular Right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Supraclavicular Left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |

LYSARC 

| Not evaluated | XX (XX.X%) |
|-------------------------|----------------|
| Axillary Right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Axillary Left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Epitrochlear Right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Epitrochlear Left | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Mediastinal | , , |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Retroperitoneal | , , |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Mesenteric | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Iliac right | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Iliac left | ( , . ) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Inguinal right | ( |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Inguinal left | 7.57 (70.5770) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |
| Other nodal involvement | ΛΛ (ΛΛ.Λ/υ) |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| 1 52 | ^^ (^^.^%) |

Listing 4.7.2-2 Other nodal involvement at baseline – Included Set (XX patients)

| | | | • |
|------------------------|------------|-------------------------|------|
| Patient identification | Inclusion | Other nodal involvement | |
| number | date | Number | Site |
| XXXXX | XX/XX/XXXX | XX | XXXX |

LYSARC 

# 5.5.3 Extra-nodal involvement

Table 4.7.3-1 Extra-nodal involvement at baseline – Included Set

| | Included Set<br>N=XX |
|----------------------------------------------------|----------------------|
| Patients with at least one extra-nodal involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Table 4.7.3-2 Description of extra-nodal involvement at baseline – Included Set

| able 4.7.3-2 | Description of extra-n | |
|---------------|------------------------|--------------|
| | | Included Set |
| | | N=XX |
| Spleen | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Liver | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Pancreas | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Pleura | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Lung | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Ascites | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Pericardium | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Breast | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Gonadal | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Kidney | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Adrenal | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Thyroid | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Skin | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |
| Soft Tissues | | |
| Normal | | XX (XX.X%) |
| Involved | | XX (XX.X%) |
| Not Evaluated | | XX (XX.X%) |

LYSARC 

| Bone | |
|-------------------------------|--------------------------|
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Blood | VV (VV V0/) |
| Normal<br>Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Tonsil | XX (XX.X%) |
| Normal | VV (VV V0/) |
| Involved | XX (XX.X%)<br>XX (XX.X%) |
| Not Evaluated | ' ' |
| Cavum | XX (XX.X%) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Parotid | XX (XX.X70) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%)<br>XX (XX.X%) |
| Orbit | ΛΛ (ΛΛ.Λ70) |
| Normal | XX (XX.X%) |
| Involved | , , , |
| Not Evaluated | XX (XX.X%)<br>XX (XX.X%) |
| | ۸۸ (۸۸.۸%) |
| Sinus<br>Normal | VV (VV V0/) |
| Involved | XX (XX.X%) |
| | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Meningeal | VV (VV V0/) |
| Normal<br>Involved | XX (XX.X%) |
| | XX (XX.X%) |
| Not Evaluated Other CNS | XX (XX.X%) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Stomach | |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Duodenum | XX (XX.X70) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Small intestine | ΛΛ (ΛΛ.Λ/0) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Ileo-caecal junction | ΛΛ (ΛΛ.Λ/0) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Colon | 701 (701.7770) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Rectum | 701 (771.7779) |
| Normal | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) |
| Other extra-nodal involvement | ΛΛ (ΛΛ.Λ/0) |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| 100 | AA (AA.A70) |

<u>Listing 4.7.3-1</u> Other extra-nodal involvement at baseline – Included Set (XX patients)

| Patient identification | Inclusion | Other extra-nodal involvement | |
|------------------------|------------|-------------------------------|------|
| number | date | Number | Site |
| XXXXX | XX/XX/XXXX | XX | XXXX |

LYSARC 

#### 5.5.4 Bone Marrow

Table 4.7.4-1 Description of BM involvement at baseline – Included Set

| | Included Set |
|----------------------|--------------|
| | N=XX |
| Bone Marrow Biopsy | |
| Not Involved | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Unspecified | XX (XX.X%) |
| Bone Marrow Aspirate | |
| Not Involved | XX (XX.X%) |
| Involved | XX (XX.X%) |
| Unspecified | XX (XX.X%) |

# 5.5.5 Staging

Table 4.7.5-1 Staging at baseline – Included Set

| | Included Set<br>N=XX |
|---------------------------|----------------------|
| Performance status (ECOG) | |
| 0 | XX (XX.X%) |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| Ann Arbor stage | |
| 1 | XX (XX.X%) |
| l II | XX (XX.X%) |
| III | XX (XX.X%) |
| IV | XX (XX.X%) |
| B symptoms | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| MIPI risk group | |
| Low risk | XX (XX.X%) |
| Intermediate risk | XX (XX.X%) |
| High risk | XX (XX.X%) |
| MIPIb risk group | |
| Low risk | XX (XX.X%) |
| Intermediate risk | XX (XX.X%) |
| High risk | XX (XX.X%) |

#### 5.5.6 MRD

Table 4.7.6-7 Informative MRD at baseline – Included Set

| Tubic 41/10 / Illioilliative Wills | at baseline int |
|--------------------------------------|-----------------|
| | Included Set |
| | N=XX |
| Patients suitable for MRD monitoring | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Baseline ddPCR Interpretation on PB | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Baseline ddPCR Interpretation on BM | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

LYSARC 

# 5.6 Evaluation during study

#### 5.6.1 Clinical examination

Table 5.6-1 Clinical examination during treatment – Safety Set

| | After Induction | After ASCT | After 3 years of | End of Treatment |
|---|---|---|---|---|
| | | | maintenance | |
| | N=XX | N=XX | N=XX | N=XX |
| Performance status (ECOG) | | | | |
| 0 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Result of Clinical Exam | | | | |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Abnormal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not done | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

#### 5.6.2 Tumor assessment

Table 5.6-2 Bone marrow results during treatment – Safety Set

| | After Induction | After ASCT | After 3 years of | End of Treatment |
|---|---|---|---|---|
| | Arter mauction | AILEI ASCI | , | End of Treatment |
| | | | maintenance | |
| | N=XX | N=XX | N=XX | N=XX |
| Bone Marrow biopsy | | | | |
| Not done | XX (XX.X%) | XX (XX.X%) | NA | XX (XX.X%) |
| Done | XX (XX.X%) | XX (XX.X%) | | XX (XX.X%) |
| If done, results: | | | | |
| Not involved | XX (XX.X%) | XX (XX.X%) | | XX (XX.X%) |
| Involved | XX (XX.X%) | XX (XX.X%) | | XX (XX.X%) |
| Unspecified | XX (XX.X%) | XX (XX.X%) | | XX (XX.X%) |
| Bone Marrow aspirate | | | | |
| Not done | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Done | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If done, results: | | | | |
| Not involved | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Involved | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Unspecified | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Listing 5.6-3 Abnormal CT scan during maintenance – Included Set (XX patients)

| Patient identification | Inclusion date | CT scan | | |
|------------------------|----------------|---------|----------|-------------|
| number | | Period | Result | Abnormality |
| XXXXX | XX/XX/XXXX | XX | Abnormal | XX |

#### 5.6.3 MRD results

Table 5.6.3-1 MRD results according to ddPCR during maintenance – Efficacy Set

| 14516 5.0.5 1 | rable 51015 1 With results according to dar cit during maintenance Lineacy Sec | | | | | |
|---|---|---|---|---|---|---|
| | During maintenance | | | | | |
| | After 6M | After 12M | 12M After 18M After 24M | | After 30M | After 36M |
| N=XX | | N=XX | N=XX | N=XX | N=XX | N=XX |
| MRD results on PB | | | | | | |
| Negative | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Table 5.6.3-2 MRD results according to ddPCR during maintenance on demand — Efficacy Set

| | | | | | | | , |
|---|---|---|---|---|---|---|---|
| | | During maintenance | | | | | |
| | After 6M After 12M | | After 18M | After 24M | After 30M | After 36M | EoT |
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| MRD results on PB | | | | | | | |
| Negative | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

LYSARC 

# **5.7 Efficacy Analysis**

# 5.7.1 Primary efficacy analysis

# 5.7.1.1 Main analysis

Table 5.7.1.1-1 MRD results on BM after induction or at treatment discontinuation – Efficacy Set

| | ddPCR | Q-PCR |
|----------------------|------------------|------------------|
| | N=XX | N=XX |
| MRD after induction | | |
| Negative | XX (XX.XX%) | XX (XX.XX%) |
| Positive | XX (XX.XX%) | XX (XX.XX%) |
| Positive < 10E-04 | XX (XX.XX%) | XX (XX.XX%) |
| Missing | XX (XX.XX%) | XX (XX.XX%) |
| MRD negativity rate* | | |
| Negative | XX (XX.XX%) | XX (XX.XX%) |
| IC 95% | [XX.XX% - XX.X%] | [XX.XX% - XX.X%] |

<sup>\*</sup> Patients without MRD assessment are considered as Positive MRD

Listing 5.7.1-1 Patients with missing MRD results on BM after induction or at treatment discontinuation – Efficacy Set (XX patients)

| Patient | Inclusion | Last period | Patient suitable for | MRD after Induction | |
|---|---|---|---|---|---|
| identification | date | | MRD monitoring | Interpretation on | Interpretation on |
| number | | | | PB | BM |
| XXXXX | XX/XX/XX | XX | XX | XX | XX |

#### 5.7.1.2 Sensitivity analysis

Table 5.7.1.21-2 MRD results on BM after induction or at treatment discontinuation – modified Efficacy Set

| | ddPCR | Q-PCR |
|---------------------|------------------|------------------|
| | N=XX | N=XX |
| MRD after induction | | |
| Negative | XX (XX.XX%) | XX (XX.XX%) |
| Positive | XX (XX.XX%) | XX (XX.XX%) |
| Positive < 10E-04 | XX (XX.XX%) | XX (XX.XX%) |
| MRD negativity rate | | |
| Negative | XX (XX.XX%) | XX (XX.XX%) |
| IC 95% | [XX.XX% - XX.X%] | [XX.XX% - XX.X%] |

LYSARC 

# 5.7.2 Progression-Free Surival (PFS)

#### 5.7.2.1 Efficacy Set

Table 5.7.2.1-1 Events according to PFS definition\* – Efficacy Set

| Table 317.212 1 Events according to 113 demini | ion Enicacy Sc |
|------------------------------------------------|----------------|
| | Efficacy Set |
| | N=XX |
| Events for PFS | |
| No event | XX (XX.X%) |
| Death without progression | XX (XX.X%) |
| Progression/relapse | XX (XX.X%) |

<sup>\*</sup> Response assessment by the investigator

Figure 5.7-1 PFS since inclusion – Efficacy Set

Table 5.7-2 PFS since inclusion – Survival Summary – Efficacy Set

| | N | Median | 95% Confidence Limits | | Min | Max |
|--------------|----|--------|-----------------------|-------|------|------|
| | | | Lower | Upper | | |
| PFS (months) | XX | XX.X | XX.X | XX.X | XX.X | XX.X |

Table 5.7-3 PFS since inclusion – Survival Estimates – Efficacy Set

| Time Point | PFS(%) | 95% Confid | 95% Confidence Limits | |
|------------|--------|------------|-----------------------|---------|
| (months) | | Lower | Upper | at risk |
| 0 | XX.X | XX.X | XX.X | XX |
| 6 | XX.X | XX.X | XX.X | XX |
| 12 | XX.X | XX.X | XX.X | XX |
| | XX.X | XX.X | XX.X | XX |

#### 5.7.2.2 Safety Set

Table 5.7-4 Events for PFS definition\* – Safety Set

| | , |
|---------------------------|------------|
| | Safety Set |
| | N=XX |
| Events for PFS | |
| No event | XX (XX.X%) |
| Death without progression | XX (XX.X%) |
| Progression/relapse | XX (XX.X%) |

<sup>\*</sup> Response assessment by the investigator

Figure 5.7-2 PFS since inclusion – Safety Set

Table 5.7-5 PFS since inclusion – Survival Summary – Safety Set

| - | | | | | | | |
|---|--------------|----|--------|-----------------------|-------|------|------|
| | | N | Median | 95% Confidence Limits | | Min | Max |
| | | | | Lower | Upper | | |
| Г | PFS (months) | XX | XX.X | XX.X | XX.X | XX.X | XX.X |

Table 5.7-6 PFS since inclusion – Survival Estimates – Safety Set

| 1 abic 3.7-0 | 1133 | mice micius | ololi July | IVAI LJUIIIC |
|--------------|--------|-------------|-----------------------|--------------|
| Time Point | PFS(%) | 95% Confid | 95% Confidence Limits | |
| (months) | | Lower | Upper | at risk |
| 0 | XX.X | XX.X | XX.X | XX |
| 6 | XX.X | XX.X | XX.X | XX |
| 12 | XX.X | XX.X | XX.X | XX |
| | XX.X | XX.X | XX.X | XX |

LYSARC 

# 5.7.3 Overall Surival (OS)

#### 5.7.3.1 Efficacy Set

Figure 5.72-2 Overall Survival – Efficacy Set

Table 5.72-4 Overall Survival – Survival Summary – Efficacy Set

| | | N | Median | 95% Confidence Limits | | Min | Max |
|---|------------|----|--------|-----------------------|-------|------|------|
| | | | | Lower | Upper | | |
| 0 | S (months) | XX | XX.X | XX.X | XX.X | XX.X | XX.X |

Table 5.72-5 Overall Survival – Survival Estimates – Efficacy Set

| Time Point | OS(%) | 95% Confidence Limits | | Patients |
|------------|-------|-----------------------|-------|----------|
| (months) | | Lower | Upper | at risk |
| 0 | XX.X | XX.X | XX.X | XX |
| 6 | XX.X | XX.X | XX.X | XX |
| 12 | XX.X | XX.X | XX.X | XX |
| | XX.X | XX.X | XX.X | XX |

#### 5.7.3.2 Safety Set

Figure 5.72-2 Overall Survival – Safety Set

Table 5.72-4 Overall Survival – Survival Summary – Safety Set

| | N | Median | 95% Confid | 95% Confidence Limits | | Max |
|-------------|----|--------|------------|-----------------------|------|------|
| | | | Lower | Upper | | |
| OS (months) | XX | XX.X | XX.X | XX.X | XX.X | XX.X |

Table 5.72-5 Overall Survival – Survival Estimates – Safety Set

| Time Point | OS(%) | 95% Confid | 95% Confidence Limits | |
|------------|-------|------------|-----------------------|---------|
| (months) | | Lower | Upper | at risk |
| 0 | XX.X | XX.X | XX.X | XX |
| 6 | XX.X | XX.X | XX.X | XX |
| 12 | XX.X | XX.X | XX.X | XX |
| | XX.X | XX.X | XX.X | XX |

# 5.7.4 Response rate

Table 5.7-6 Response according to Cheson 99 – Efficacy Set

| | Evaluation after 3 years | End of treatment |
|-------------------------------|--------------------------|------------------|
| | of maintenance | |
| | N=XX | N=XX |
| Response (Cheson 99) | | |
| Complete Metabolic Response | XX (XX.X%) | XX (XX.X%) |
| Partial Metabolic Response | XX (XX.X%) | XX (XX.X%) |
| No Metabolic Response | XX (XX.X%) | XX (XX.X%) |
| Progressive Metabolic Disease | XX (XX.X%) | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) | XX (XX.X%) |
| Overall Response Rate (ORR) | | |
| Patients with ORR | XX (XX.X%) | XX (XX.X%) |
| IC 95% | [XX.X% - XX.X%] | [XX.X% - XX.X%] |
| Overall Response Rate* (ORR) | | |
| Patients with ORR | XX (XX.X%) | XX (XX.X%) |
| IC 95% | [XX.X% - XX.X%] | [XX.X% - XX.X%] |

<sup>\*</sup> Patients who relapsed or died during treatment phase are considered as non-responders even if they were repsonders before withdrawal.

LYSARC 

Table 5.7-2 Response according to Cheson 99 – Safety Set

| | Evaluation after 3 years | End of treatment |
|-------------------------------|--------------------------|------------------|
| | of maintenance | |
| | N=XX | N=XX |
| Response (Cheson 99) | | |
| Complete Metabolic Response | XX (XX.X%) | XX (XX.X%) |
| Partial Metabolic Response | XX (XX.X%) | XX (XX.X%) |
| No Metabolic Response | XX (XX.X%) | XX (XX.X%) |
| Progressive Metabolic Disease | XX (XX.X%) | XX (XX.X%) |
| Not Evaluated | XX (XX.X%) | XX (XX.X%) |
| Overall Response Rate (ORR) | | |
| Patients with ORR | XX (XX.X%) | XX (XX.X%) |
| IC 95% | [XX.X% - XX.X%] | [XX.X% - XX.X%] |
| Overall Response Rate* (ORR) | | |
| Patients with ORR | XX (XX.X%) | XX (XX.X%) |
| IC 95% | [XX.X% - XX.X%] | [XX.X% - XX.X%] |

<sup>\*</sup> Patients who relapsed or died during treatment phase are considered as non-responders even if they were repsonders before withdrawal.

# 5.7.5 PET results

Table 5.7-7 PET scan result – Efficacy Set

| | After Induction | After ASCT | After 3 years of | End of Treatment |
|---|---|---|---|---|
| | /cduction | , iiici Asci | maintenance | 2.1.a or redunient |
| | N=XX | N=XX | N=XX | N=XX |
| PET scan | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If done, hypermetabolic lesion | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If yes, SUV Max tumoral | | | | |
| N | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1 ; Q3 | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX |
| If yes, localisation | | | | |
| XXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Table 5.7-2 PET scan result – Safety Set

| | After Induction | After ASCT | After 3 years of | End of Treatment |
|---|---|---|---|---|
| | | | maintenance | |
| | N=XX | N=XX | N=XX | N=XX |
| PET scan | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If done, hypermetabolic lesion | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If yes, SUV Max tumoral | | | | |
| N | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1 ; Q3 | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX |
| If yes, localisation | | | | |
| XXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

LYSARC 

#### 5.7.6 MRD results

Table 5.7.6-1 MRD results according to ddPCR on BM – Efficacy Set

| | After 36M of | After 36M of | End of treatment |
|-------------------|--------------|-----------------------|------------------|
| | maintenance | maintenance on-demand | |
| | N=XX | N=XX | N=XX |
| MRD results on BM | | | |
| Negative | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

# 5.7.7 Duration of MRD negativity

Table 5.7.7 Events since first MRD negativity – Efficacy Set

| | Efficacy Set |
|--------------------------------------------|--------------|
| | N=XX |
| Patients with MRD negativity | XX |
| If yes, time to first negative MRD | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX ; XX |
| Min ; Max | XX ; XX |
| Event according to MRD negativity duration | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Duration of MRD negativity is defined as the time from the date of attainment the first negative MRD to the date of positive MRD. For patients achieving a negative MRD but who have not positive MRD or not MRD assessment at the time of analysis, duration of MRD negativity will be censored on the date of last MRD assessment.

Figure 5.7.7 Duration of MRD negativity – Efficacy Set

Table 5.7.7 Duration of MRD negativity – Efficacy Set – Survival Estimates

#### 5.7.8 Stem cell collection failure

Table 5.7.3.2-1 Description of stem cell collection failure – Safety Set

| | Safety Set |
|--------------------------------------|--------------|
| | , |
| | N=XX |
| Leukapheresis | |
| Done | XX (XX.X%) |
| Not Done | XX (XX.X%) |
| If not done, specify the reason: | |
| Progression | XX (XX.X%) |
| Collection failure | XX (XX.X%) |
| Toxicity | XX (XX.X%) |
| Other | XX |
| If collection failure, specify: | |
| Sepsis | XX (XX.X%) |
| Not enough cells | XX (XX.X%) |
| Logistical problem | XX (XX.X%) |
| Other cause | XX |
| If done, Total collected cells CD34+ | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1 ; Q3 | XX;XX |
| Min ; Max | XX;XX |

LYSARC 

# 5.8 Progression / Relapse

Table 5.88-1 Summary of progression/relapse – Safety Set

| | , |
|---------------------------------------|--------------|
| | Safety Set |
| | N=XX |
| Patients who progressed/relapsed | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, time since inclusion (months) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

Table 5.88-2 Involvement at progression/relapse – Safety Set

| | . 06. coo.o, . c.apoc oa |
|-------------------------|--------------------------|
| | Safety Set |
| | N=XX |
| Progression/Relapse | XX |
| Initial Involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| New Involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Nodal Involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Extra-nodal Involvement | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Table 5.88-3 Treatment for progression/relapse – Safety Set

| | Safety Set |
|-------------------------------|------------|
| | N=XX |
| Progression/relapse | XX |
| Progression/relapse treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, | |
| Monoclonal antibody | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Other immunotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Ibrutinib | |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |
| Chemotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Radiotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Autologous transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Allogenic transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, allograft transplant | |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |
| IMiD | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

LYSARC 
| Epigenetic modifiers agents | |
|-----------------------------|------------|
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Kinase inhibitor | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Other anti-cancer therapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

### Listing 5.88-1 Patients who received chemotherapy for progression/relapse – Safety Set (XX patients)

| Patient | Inclusion | Date of | Treatment for progression | | |
|---|---|---|---|---|---|
| identification | date | progression | Chemotherapy | Date | Description |
| number | | | | | |
| XXXXX | XX/XX/XX | XX/XX/XXXX | Yes | XX/XX/XXXX | XXX |

Same listing for other treatment received by at least 1 patient (no listing will be provided if empty):

- Radiotherapy
- Monoclonal Antibody
- \_

Table 5.88-4 Response according to Cheson 99 after treatment for progression/relapse – Safety Set

| | Safety Set |
|-------------------------------|------------|
| | N=XX |
| Progression/relapse | XX |
| Response | |
| Complete response | XX (XX.X%) |
| Unconfirmed complete response | XX (XX.X%) |
| Partial response | XX (XX.X%) |
| Stable disease | XX (XX.X%) |
| Progressive disease | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |

LYSARC 

## 5.9 Extent of exposure

### **5.9.1** Cycles

Table 5.9-1 Cycles perfomed – Safety set

| | Safety set |
|-----------------|------------|
| | N=XX |
| Cycle performed | |
| Cycle 1 | XX (XX.X%) |
| Cycle 2 | XX (XX.X%) |
| Cycle 3 | XX (XX.X%) |
| Cycle 4 | XX (XX.X%) |

Table 5.9-2 Number of cycles perfored – Safety set

| | Safety set |
|----------------------------|--------------|
| | N=XX |
| Number of cycles performed | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

Table 5.99.1-3 Treatment intake duration – Safety set

| | Safety set |
|------------------------------------|--------------|
| | N=XX |
| Treatment intake duration (months) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |

Treatment intake duration is defined as the time between the 1st intake of any induction drugs and the last intake of any induction drugs.

LYSARC 

#### 5.9.2 Dose

Table 5.9-3 GA101 administration by cycle during induction period – Safety set

| | | Cycle 1 | | Cycle 2 | Cycle 3 | Cycle 4 |
|---|---|---|---|---|---|---|
| | Day 1 | Day 8 | Day 15 | Day 1 | Day 1 | Day 1 |
| | N=XX | N=XX | N=XX | N=XX | N=XX | N=XX |
| Total dose taken (mg/m²) | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1; Q3 | XX;XX | XX ; XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX ; XX | XX;XX | XX;XX | XX;XX | XX;XX |
| PPD (%) | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1; Q3 | XX;XX | XX ; XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX ; XX | XX;XX | XX;XX | XX;XX | XX;XX |
| PPD (%) | | | | | | |
| < 75% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| [75% - 90%] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| [90% - 110%] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| [110% - 125%] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| >= 125% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Expected dose per cycle for GA101: 1000mg D1 + 1000mg D8 + 1000mg D15 of cycle 1.

Total dose is the sum of dose administered during one day of a cycle.

PPD = (Total dose taken/total dose expected)/100

Table 5.9-2 GA101 administration during induction period – Safety set

| | Safety set |
|--------------------------|--------------|
| | N=XX |
| Total dose taken (mg/m²) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1 ; Q3 | XX ; XX |
| Min ; Max | XX ; XX |
| PPD (%) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| PPD (%) | |
| < 75% | XX (XX.X%) |
| [75% - 90%] | XX (XX.X%) |
| [90% - 110%] | XX (XX.X%) |
| [110% - 125%] | XX (XX.X%) |
| >= 125% | XX (XX.X%) |

Expected total dose during induction for GA101 : 6000mg.

Total dose is the sum of dose administered during induction.

PPD = (Total dose taken/total dose expected)/100

LYSARC 

Table 5.9-3 GA101 administration during ASCT – Safety set

| | Safety set |
|--------------------------|--------------|
| | N=XX |
| Total dose taken (mg/m²) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1 ; Q3 | XX;XX |
| Min ; Max | XX;XX |
| PPD (%) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1 ; Q3 | XX;XX |
| Min ; Max | XX;XX |
| PPD (%) | |
| < 75% | XX (XX.X%) |
| [75% - 90%] | XX (XX.X%) |
| [90% - 110%] | XX (XX.X%) |
| [110% - 125%] | XX (XX.X%) |
| >= 125% | XX (XX.X%) |

Expected total dose during asct for GA101: 1000mg.

Total dose is the sum of dose administered during asct.

PPD = (Total dose taken/total dose expected)/100

Table 5.9-4 GA101 administration during maintenance – Safety set

| | Safety set |
|--------------------------|--------------|
| | N=XX |
| Total dose taken (mg/m²) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| PPD (%) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |
| PPD (%) | |
| < 75% | XX (XX.X%) |
| [75% - 90%] | XX (XX.X%) |
| [90% - 110%] | XX (XX.X%) |
| [110% - 125%] | XX (XX.X%) |
| >= 125% | XX (XX.X%) |

Expected total dose during maintenance for GA101: 1000mg every 2 months.

Total dose is the sum of dose administered during maintenance.

PPD = (Total dose taken/total dose expected)/100

LYSARC 

Table 5.9-5 GA101 administration during maintenance on-demand – Safety set

| | Safety set |
|--------------------------|--------------|
| | N=XX |
| Total dose taken (mg/m²) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1 ; Q3 | XX;XX |
| Min ; Max | XX;XX |
| PPD (%) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX ; XX |
| PPD (%) | |
| < 75% | XX (XX.X%) |
| [75% - 90%] | XX (XX.X%) |
| [90% - 110%] | XX (XX.X%) |
| [110% - 125%] | XX (XX.X%) |
| >= 125% | XX (XX.X%) |

Expected total dose during maintenance for GA101 if positive MRD: 3000mg for the 1st month and then 1000mg every month.

Total dose is the sum of dose administered during maintenance on-demand.

PPD = (Total dose taken/total dose expected)/100

Table 5.9-6 Patients with at least one dose interruption of GA101 – Safety set

| | Safety set |
|-------------------------------------------------------|------------|
| | N=XX |
| Patients with at least one dose interruption of GA101 | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

Listing 5.9-1 Patients with at least one dose interruption of GA101 – Safety set (XX patients)

| Patient | | Number of | | | A | Adverse Event | | |
|---|---|---|---|---|---|---|---|---|
| identification | Inclusion date | Number of | Period | Descritption | Highest | Relationship with | Action taken | Outcome |
| number | | cycles received | | | grade | GA101 | on GA101 | |
| XXXXX | XX/XX/XXXX | XX | XX | XX | Χ | XX | XX | XX |

Filter: Action taken on GA101 = Drug interrupted

LYSARC 

## **5.10** Safety analysis

### **5.10.1** Adverse Events

Table 5.101-1 Summary of AEs – Safety set

| | Induction | ASCT | Maintenance | Total |
|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX |
| Patients with at least one AE | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If yes, number of Aes by patients | | | | |
| N | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1;Q3 | XX;XX | XX;XX | XX;XX | XX ; XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX ; XX |
| Patient with at least one AE of grade >= 3 | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Patient with at least one fatal AE | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Patient with at least one AE leading to treatment discontinuation | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Patient with at least one AESI* | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>\*</sup> AESI = Tumor Lysis Syndrom and IRR grade 4 occuring during or within 24 hours after the GA101 infusion.

Table 5.101-2 Summary of related AEs – Safety set

| | Induction | ASCT | Maintenance | Total |
|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX |
| Patients with at least one related AE | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If yes, number of related Aes by patients | | | | |
| N | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1;Q3 | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX |
| Patient with at least one related AE of grade >= 3 | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Patient with at least one fatal related AE | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Patient with at least one related AE leading to treatment discontinuation | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Patient with at least one related AESI* | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>\*</sup> AESI = Tumor Lysis Syndrom and IRR grade 4 occurring during or within 24 hours after the GA101 infusion.

LYSARC 

Table 5.101-3 AEs by SOC and PT – Safety set

| Safety set |
|------------|
| N=XX |
| XX (XX.X%) |
| XX (XX.X%) |
| XX (XX.X%) |
| XX (XX.X%) |
| XX (XX.X%) |
| XX (XX.X%) |
| XX (XX.X%) |

Table 5.101-4 Description of AEs by SOC/PT and by highest intensity – Safety set

| System Organ Class | Gra | de 3 | Gra | de 4 | Grade 5 | |
|---|---|---|---|---|---|---|
| | N= | :XX | N= | :XX | N=XX | |
| Preferred Term | Patients | Events | Patients | Events | Patients | Events |
| AEs | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SOC 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PT 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PT | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SOC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PT 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PT | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Table 5.101-5 Characteristics of AEs – Safety set

| able 5.101-5 Characteristics of AE | Safety set |
|------------------------------------|------------|
| | N=XX |
| Onset period | |
| Before pr-phase | XX (XX.X%) |
| Pre-phase | XX (XX.X%) |
| Induction | XX (XX.X%) |
| ASCT | XX (XX.X%) |
| Maintenance | XX (XX.X%) |
| Maintenance on-demand | XX (XX.X%) |
| Follow-up | XX (XX.X%) |
| Highest intensity | |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| Relationship with GA101 | |
| Unrelated | XX (XX.X%) |
| Related | XX (XX.X%) |
| Not applicable | XX (XX.X%) |
| Relationship with DHAP | |
| Unrelated | XX (XX.X%) |
| Related | XX (XX.X%) |
| Not applicable | XX (XX.X%) |
| Relationship with ASCT | |
| Unrelated | XX (XX.X%) |
| Related | XX (XX.X%) |
| Not applicable | XX (XX.X%) |
| Serious AE | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| AESI* | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Outcome | |
| Not recovered/Not resolved | XX (XX.X%) |
| Recovered/Resolved | XX (XX.X%) |
| Recovered/Resolved with sequelae | XX (XX.X%) |
| Recovering/Resolving | XX (XX.X%) |
| Fatal | XX (XX.X%) |

<sup>\*</sup> AESI = Tumor Lysis Syndrom and IRR grade 4 occuring during or within 24 hours after the GA101 infusion.

LYSARC 

Listing 5.10.1-1 Patients with fatal AEs – Safety set (XX AEs reported by XX patients)

| Patient | Inclusion | Number | | | | P | Adverse Event | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| identification | date | of | | | | Event | Date when | Highest | GA101 | | Outcome |
| number | | cycles | Number | Description | Onset date | period | AE became | intensity | Relationship | Action | |
| | | received | | | | | serious | intensity | | taken | |
| XXXXX | XX/XX/XXXX | Χ | Yes | XXXXX | XX/XX/XXXX | XX | XX/XX/XXXX | Χ | X | XX | XXX |

## Listing 5.10.1-2 Patients with AEs leading to treatment discontinuation – Safety set (XX AEs reported by XX patients)

| Patient | Inclusion | Number | Adverse Event | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| identification | date | of | | | | Event | Date when | Highest | GA101 | | Outcome |
| number | | cycles | Number | Description | Onset date | period | AE became | intensity | Relationship | Action | |
| | | received | | | | | serious | intensity | | taken | |
| XXXXX | XX/XX/XXXX | Х | Yes | XXXXX | XX/XX/XXXX | XX | XX/XX/XXXX | Х | Х | XX | XXX |

Listing 5.10.1-3 Patients with AESI\* – Safety set (XX AEs reported by XX patients)

| Patient | Inclusion | Number | | | | F | Adverse Event | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| identification | date | of | | | | Event | Date when | Highest | GA101 | L | Outcome |
| number | | cycles | Number | Description | Onset date | period | AE became | intensity | Relationship | Action | |
| | | received | | | | | serious | intensity | | taken | |
| XXXXX | XX/XX/XXXX | X | Yes | XXXXX | XX/XX/XXXX | XX | XX/XX/XXXX | Х | X | XX | XXX |

<sup>\*</sup> AESI = Tumor Lysis Syndrom and IRR grade 4 occuring during or within 24 hours after the GA101 infusion

### **5.10.2** Serious Adverse Events

Table 5.102-2 Summary of SAEs - Safety set

| Table 5.102-2 Summary of SAES – Safety Set | |
|---------------------------------------------|------------|
| | Safety set |
| | N=XX |
| Patients with at least one SAE | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Patient with at least one related SAE | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Patient with at least one SAE of grade >= 3 | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

#### Table 5.102-3 SAEs by SOC and PT – Safety set

| . 45.0 5.202 5 | or izo by occurrent oursely see |
|----------------|---------------------------------|
| | Safety set |
| | N=XX |
| AEs | XX (XX.X%) |
| SOC 1 | XX (XX.X%) |
| PT 1 | XX (XX.X%) |
| PT | XX (XX.X%) |
| SOC | XX (XX.X%) |
| PT 1 | XX (XX.X%) |
| PT | XX (XX.X%) |

#### Table 5.102-3 Related SAEs by SOC and PT – Safety set

| 1 able 2.102-3 | Related SAES by SOC allu P | ı – Saiety set |
|----------------|----------------------------|----------------|
| | | Safety set |
| | | N=XX |
| Related SAEs | | XX (XX.X%) |
| SOC 1 | | XX (XX.X%) |
| PT 1 | | XX (XX.X%) |
| PT | | XX (XX.X%) |
| SOC | | XX (XX.X%) |
| PT 1 | | XX (XX.X%) |
| PT | | XX (XX.X%) |

LYSARC 

Table 5.102-4 Characteristics of SAEs – Safety set

| Table 5.102-4 Characteristics of SAEs – Safety set | |
|----------------------------------------------------|------------|
| | Safety set |
| | N=XX |
| Onset period | |
| Pre-phase | XX (XX.X%) |
| Induction | XX (XX.X%) |
| ASCT | XX (XX.X%) |
| Maintenance | XX (XX.X%) |
| Maintenance on-demand | XX (XX.X%) |
| Follow-up | XX (XX.X%) |
| Highest intensity | |
| 1 | XX (XX.X%) |
| 2 | XX (XX.X%) |
| 3 | XX (XX.X%) |
| 4 | XX (XX.X%) |
| 5 | XX (XX.X%) |
| Relationship with GA101 | |
| Unrelated | XX (XX.X%) |
| Related | XX (XX.X%) |
| Not applicable | XX (XX.X%) |
| Relationship with DHAP | |
| Unrelated | XX (XX.X%) |
| Related | XX (XX.X%) |
| Not applicable | XX (XX.X%) |
| Relationship with ASCT | |
| Unrelated | XX (XX.X%) |
| Related | XX (XX.X%) |
| Not applicable | XX (XX.X%) |
| Serious AE | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| AESI* | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Outcome | |
| Not recovered/Not resolved | XX (XX.X%) |
| Recovered/Resolved | XX (XX.X%) |
| Recovered/Resolved with sequelae | XX (XX.X%) |
| Recovering/Resolving | XX (XX.X%) |
| Fatal | XX (XX.X%) |

<sup>\*</sup> AESI = Tumor Lysis Syndrom and IRR grade 4 occurring during or within 24 hours after the GA101 infusion

Listing 5.10.2-2 Patients with SAEs – Safety set (XX SAEs reported by XX patients)

| Patient | Inclusion | Number | | Adverse Event | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| identification | date | of | | | | Event | Date when | Highest | GA101 | L | Outcome |
| number | | cycles | Number | Description | Onset date | period | AE became | intensity | Relationship | Action | |
| | | received | | | | | serious | intensity | | taken | |
| XXXXX | XX/XX/XXXX | X | Yes | XXXXX | XX/XX/XXXX | XX | XX/XX/XXXX | Х | X | XX | XXX |

LYSARC 

### 5.10.3 Other Primay Malignancy (OPM)

Table 5.10.4 OPM – Safety set

| | Safety set |
|-----------------------------------------------------------|--------------|
| | N=XX |
| Patients with at least one OPM | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, number of OPMs by patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| If yes, time to onset of 1st OPM since inclusion (months) | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX;XX |

### Table 5.10-5 OPM by SOC and PT – Safety set

| | Safety | set |
|-------|------------|--------|
| | N=X | (X |
| | Patients | Events |
| ОРМ | XX (XX.X%) | XX |
| SOC 1 | XX (XX.X%) | XX |
| PT 1 | XX (XX.X%) | XX |
| PT | XX (XX.X%) | XX |
| SOC | XX (XX.X%) | XX |
| PT 1 | XX (XX.X%) | XX |
| PT | XX (XX.X%) | XX |

### Listing 5.10-1 OPM – Safety set (XX patients)

| Patient | Inclusion | | OPM | | | | Death | Study |
|---|---|---|---|---|---|---|---|---|
| identification<br>number | date | Date | Time since inclusion (months) | Description | Y/N | Cause | Other concurrent illness description | duration<br>(months) |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX | XXX | XX | XXX | XXX | XXX |

Listing 5.10-2 Narratives of OPMs – Safety set (XX patients)

| Patient identification | Inclusion | OPM | | |
|---|---|---|---|---|
| number | date | Date | Description | Narrative |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX | XX |

LYSARC 

### 5.10.4 Deaths

Table 5.10-6 Deaths – Safety set

| | Safety set<br>N=XX |
|--------------------------------------------------------|--------------------|
| Death | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, cause of death | |
| Lymphoma | XX (XX.X%) |
| Toxicity of study treatment (including related cancer) | XX (XX.X%) |
| Concurrent illness | XX (XX.X%) |
| Toxicity of additional treatment | XX (XX.X%) |
| Other cause | XX (XX.X%) |
| Unknown | XX (XX.X%) |
| If yes, phase of death | |
| Induction phase | XX (XX.X%) |
| ASCT | XX (XX.X%) |
| Maintenance phase | XX (XX.X%) |
| Follow-Up | XX (XX.X%) |
| Disease status at death | |
| Complete response | XX (XX.X%) |
| Unconfirmed Complete response | XX (XX.X%) |
| Partial response | XX (XX.X%) |
| Stable disease | XX (XX.X%) |
| Progressive disease | XX (XX.X%) |
| Not evaluated | XX (XX.X%) |

Listing 5.10.4-3 Deaths – Safety set (XX patients)

| | | | ( | , | | | | |
|---|---|---|---|---|---|---|---|---|
| Patient | Inclusion | Number of | Study | | | Deat | :h | |
| identification | date | cvcles | duration | Date | Cause | Specification of | Specification of | Specification of |
| number | | received | (months) | | | concurrent | other concurrent | other reason |
| | | receiveu | (IIIOIILIIS) | | | illness | illness | |
| XXXXX | XX/XX/XXXX | Х | XX.X | XX/XX/XXXX | XXXXX | XXXXX | XXXXX | XXXXX |

Listing 5.10.4-4 Narratives of fatal SAE – Safety set (XX patients)

| Patient identification | Inclusion | OPM | | |
|---|---|---|---|---|
| number | date | Date | Description | Narrative |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX | XX |

LYSARC 

## 5.10.5 Clinical Laboratory

Table 5.10-7 Hematology from baseline to End of Treatment – Safety set

| | Baseline | End of | ASCT | After 3y of | EoT |
|---|---|---|---|---|---|
| | | induction | | maintenance | |
| | N=XX | N=XX | N=XX | N=XX | N=XX |
| Hematology done | | | | | |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If yes, | | | | | |
| Hemoglobin (g/dL) | | | | | |
| N | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1 ; Q3 | XX;XX | XX ; XX | XX;XX | XX ; XX | XX ; XX |
| Min ; Max | XX;XX | XX ; XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX ; XX | XX ; XX | XX;XX |
| Leukocytes (g/L) | | | | | |
| N | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1 ; Q3 | XX;XX | XX ; XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX ; XX | XX;XX | XX ; XX | XX;XX |
| Min ; Max | XX;XX | XX ; XX | XX;XX | XX;XX | XX;XX |
| Neutrophils (g/L) | | | | | |
| N | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1;Q3 | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Lymphocytes (g/L) | | | | | |
| N | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1;Q3 | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Presence of lymphoma cells (g/L) | | | | | |
| N | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1 ; Q3 | XX;XX | XX ; XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Platelets (g/L) | | | | | |
| N | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1; Q3 | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |
| Min ; Max | XX;XX | XX;XX | XX;XX | XX;XX | XX;XX |

LYSARC 

Table 5.10-2 Biochemistry from baseline to ASCT – Safety set

| Median XX, X XX, X XX, X XX, X XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX <t< th=""><th>Table 5.10-2 Biochemistry from</th><th>paseline to A</th><th>SCT – Safety set</th><th></th></t<> | Table 5.10-2 Biochemistry from | paseline to A | SCT – Safety set | |
|---|---|---|---|---|
| Biochemistry done | | Baseline | End of induction | ASCT |
| No | | N=XX | N=XX | N=XX |
| Yes | Biochemistry done | | | |
| Yes | | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| If yes, AST (IU/L) N | | , , , | | |
| AST (IU/L) XX | | | (, | ( , . , |
| N XX XX XX XX XX XX XX | • • | | | |
| Missing Mean (SD) XX XXX | | VY | VY. | VY |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) <td></td> <td></td> <td></td> <td></td> | | | | |
| Median XX.X | _ | | | |
| Q1; Q3 XX; XX XX | ļ , , | 1 ' | | |
| Min; Max XX; XX XX XX< | | | | |
| Min Max | | | | |
| ALT (IU/L) N | , | | | · · |
| N N N N N XX XX XX XX | | XX;XX | XX;XX | XX;XX |
| Missing | , , , | | | |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) <td></td> <td></td> <td></td> <td></td> | | | | |
| Median XX.X | Missing | XX | XX | |
| Q1; Q3 | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Min; Max Min; Max Min; Max Min; Max XX; XX XX | Median | XX.X | XX.X | XX.X |
| Min ; Max | Q1; Q3 | XX;XX | XX;XX | XX ; XX |
| Total bilirubin (μmol/L) | Min ; Max | XX;XX | XX;XX | XX;XX |
| N | Min ; Max | XX;XX | XX ; XX | XX ; XX |
| N | Total bilirubin (µmol/L) | | | |
| Missing Mean (SD) XX XX XX XX XX.X (XX.XX) XX.X (XX.XX XX.X (XX.XX) | | XX | xx | xx |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) <td></td> <td></td> <td></td> <td></td> | | | | |
| Median XX.X | _ | | | |
| Q1; Q3 XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX <td>, ,</td> <td>1 '</td> <td></td> <td></td> | , , | 1 ' | | |
| Min; Max XX; XX XX | | | | |
| Min; Max | | | | |
| Serum creatinine (μmol/L) N XX XX XX XX XX XX XX | - | 1 | | |
| N XX XX< | - | ^^,^^ | ^^,^^ | ^^,^^ |
| Missing Mean (SD) XX | | | | |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) <td></td> <td></td> <td></td> <td></td> | | | | |
| Median XX.X | _ | | | |
| Q1; Q3 XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX <t< td=""><td>ļ , ,</td><td>, ,</td><td>, , ,</td><td></td></t<> | ļ , , | , , | , , , | |
| Min; Max XX; XX XX | | | | |
| Min; Max XX; XX XX; XX XX; XX Creatinine clearance Cockcroft-Gault formula (μmol/L) XX < | | | | |
| Creatinine clearance Cockcroft-Gault formula (μmol/L) XX XX< | | | | |
| Cockcroft-Gault formula (μmol/L) N XX | · | XX ; XX | XX ; XX | XX ; XX |
| N XX XX< | Creatinine clearance | | | |
| Missing XX XX XX XX XX.X (XX.XX) < | Cockcroft-Gault formula (μmol/L) | | | |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) <td>N</td> <td>XX</td> <td>XX</td> <td>XX</td> | N | XX | XX | XX |
| Median XX.X | Missing | XX | XX | XX |
| Q1; Q3 XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX <t< td=""><td>Mean (SD)</td><td>XX.X (XX.XX)</td><td>XX.X (XX.XX)</td><td>XX.X (XX.XX)</td></t<> | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Q1; Q3 XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX; XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX <t< td=""><td></td><td></td><td></td><td></td></t<> | | | | |
| Min; Max XX; XX XX | Q1;Q3 | XX;XX | XX;XX | XX;XX |
| Min; Max XX; XX XX; XX XX; XX MDRD formula (μmol/L) XX XX XX XX Missing XX | Min ; Max | XX;XX | XX;XX | XX;XX |
| MDRD formula (μmol/L) XX XX< | | | | |
| N XX XX< | | , | , | , |
| Missing XX XX XX XX XX.X (XX.XX) < | | XX | XX | XX |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) <td></td> <td></td> <td></td> <td></td> | | | | |
| Median XX.X | | | | |
| Q1; Q3 XX; XX XX | ` ' | 1 ' | , , | |
| Min; Max XX; XX XX | | | | |
| Min; Max XX; XX XX; XX XX; XX CKD-EPI formula (μmol/L) XX XX XX N Missing XX XX XX Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X XX.X Q1; Q3 XX; XX XX; XX XX; XX | · · | | | · · |
| CKD-EPI formula (μmol/L) N XX XX XX Missing XX XX XX Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X XX.X Q1; Q3 XX; XX XX; XX XX; XX | | | | |
| N XX XX XX Missing XX XX XX Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X XX.X Q1; Q3 XX; XX XX; XX XX; XX | | ^^; ^^ | ^^;^^ | ^^; ^^ |
| Missing XX XX XX Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X XX.X Q1; Q3 XX; XX XX; XX XX; XX | " , , | ,,,, | , | \ \. |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) Median XX.X XX.X XX.X Q1; Q3 XX; XX XX; XX XX; XX | | | | |
| Median XX.X XX.X XX.X Q1; Q3 XX; XX XX; XX XX; XX | | | | |
| Q1; Q3 | | 1 ' | | XX.X (XX.XX) |
| Min · May | · · | | | |
| | Min ; Max | XX ; XX | XX ; XX | XX ; XX |
| Min ; Max XX ; XX XX ; XX XX ; XX | Min ; Max | XX;XX | XX ; XX | XX ; XX |

LYSARC 

### **5.11** Concomitant treatments

#### 5.11.1 Concomitant treatments at inclusion

Table 5.11-1 Concomitant treatments before baseline\* – Included Set

| | Included Set |
|---------------------------------------------------------|--------------|
| | N=XX |
| Patients with at least one concomitant treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, number of concomitant treatment per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Patients with at least one concomitant treatment due to | |
| lymphoma | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

<sup>\*</sup> Concomitant treatment started before C1D1 and ended before C1D1.

Listing 5.11-1 Concomitant treatments before baseline\* – Included Set (XX patients)

| Patient | Inclusion | C1D1 | Concomitant treatment | | | | | |
|---|---|---|---|---|---|---|---|---|
| identification | date | | Start date | Number | Drug Name | Indication | End date | Ongoing |
| number | | | | | (INN) | | | |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX/XX/XXXX | XX | XXX | XX | XX/XX/XXXX | Х |

<sup>\*</sup> Concomitant treatment started before C1D1 and ended before C1D1.

Table 5.11-2 Concomitant treatments at baseline\* – Included Set

| | Included Set |
|---------------------------------------------------------|--------------|
| | N=XX |
| Patients with at least one concomitant treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, number of concomitant treatment per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1 ; Q3 | XX;XX |
| Min ; Max | XX;XX |
| Patients with at least one concomitant treatment due to | |
| lymphoma | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

<sup>\*</sup> Concomitant treatment started before C1D1 and ended during treatment or still on going.

Listing 5.11-2 Concomitant treatments at baseline\* – Included Set (XX patients)

| Patient | Inclusion | C1D1 | Concomitant treatment | | | | | |
|---|---|---|---|---|---|---|---|---|
| identification | date | | Start date | Indication | End date | Ongoing | | |
| number | | | | | (INN) | | | |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX/XX/XXXX | XX | XXX | XX | XX/XX/XXXX | Х |

<sup>\*</sup> Concomitant treatment started before C1D1 and ended during treatment or still on going.

LYSARC 

### 5.11.2 Concomitant treatments during treatment period

Table 5.112-2 Concomitant treatments during treatment\* – Included Set

| | Included Set |
|---------------------------------------------------------|--------------|
| | N=XX |
| Patients with at least one concomitant treatment | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, number of concomitant treatment per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1; Q3 | XX ; XX |
| Min ; Max | XX ; XX |
| Patients with at least one concomitant treatment due to | |
| lymphoma | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

<sup>\*</sup> Concomitant treatment started after C1D1 or with missing starting dates but still on going.

Listing 5.112-2 Concomitant treatments during treatment\* – Included Set (XX patients)

| Patient | Inclusion | C1D1 | Concomitant treatment | | | | | |
|---|---|---|---|---|---|---|---|---|
| identification | date | | Start date Number Drug Name Indication End date Ongoin | | | | | |
| number | | | | | (INN) | | | |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX/XX/XXXX | XX | XXX | XX | XX/XX/XXXX | Х |

<sup>\*</sup> Concomitant treatment started after C1D1 or with missing starting dates but still on going.

### 5.12 Non study treatments out of progression

Table 5.122-1 Non study treatment treatment out of progression – Safety Set

| | Safety Set |
|----------------------------------------|------------|
| | N=XX |
| Non study treatment out of progression | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Monoclonal antibody | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Other immunotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Chemotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Radiotherapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Autologous transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Allogenic transplant | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, IMiD | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Epigenetic modifiers agents | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Kinase inhibitors | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, Other anti-cancer therapy | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |

LYSARC 

## Listing 5.122-1 Patients who received monoclonal antibody as non study treatment treatment out of progression – Safety Set (XX patients)

| Patient | Inclusion | Permanent treatment | | Non study treatment treatment out of progression | | |
|---|---|---|---|---|---|---|
| identification | date | discontinuation | | | | |
| number | | Date Reason | | Monoclonal | Date | Drug name |
| | | | | antibody | | |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX | Yes | XX/XX/XXXX | XXX |

## Listing 5.122-2 Patients who received other immunotherapy as non study treatment treatment out of progression – Safety Set (XX patients)

| p 6 | ty cot (sat pane | , | | | | |
|---|---|---|---|---|---|---|
| Patient | Inclusion | Permanent | treatment | Non study treatment treatment out of progression | | |
| identification | date | discontinuation | | | | |
| number | | Date Reason | | Other | Date | Drug name |
| | | | | immunotherapy | | |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX | Yes | XX/XX/XXXX | XXX |

## Listing 5.122-3 Patients who received chemotherapy as non study treatment treatment out of progression – Safety Set (XX patients)

| Patient | Inclusion | Permanen | t treatment | Non study treatment treatment out of progression | | |
|---|---|---|---|---|---|---|
| identification | date | discontinuation | | | | |
| number | | Date | Date Reason | | Date | Drug name |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX | Yes | XX/XX/XXXX | XXX |

## Listing 5.122-4 Patients who received autologous transplant as non study treatment treatment out of progression – Safety Set (XX patients)

| P. 08. 000.0 | rogression surety see (70) patients | | | | | | |
|---|---|---|---|---|---|---|---|
| Patient | Inclusion | Permanent tr | eatment | No | Non study treatment treatment out of progression | | |
| identification | date | discontinu | ation | | | | |
| number | | Date | Reason | Autologous | Date of | Type of autologous | Date of |
| | | | | transplant | transplant | transplant intensive | autologous |
| | | | | | | chemotherapy with | transplant |
| | | | | | | HSCT | intensive |
| | | | | | | | chemotherapy |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX | Yes | XX/XX/XXXX | XXX | XX/XX/XXXX |

## Listing 5.122-5 Patients who received allogenic transplant as non study treatment treatment out of progression – Safety Set (XX patients)

| P. 05. C33.011 | Togression Surety Set (Art putients) | | | | | | |
|---|---|---|---|---|---|---|---|
| Patient | Inclusion | Permanent tr | eatment | N | Non study treatment treatment out of progression | | |
| identification | date | discontinu | ation | | | | |
| number | | Date | Reason | Allogenic | Date of | Type of allogenic | Date of allogenic |
| | | | | transplant | transplant | transplant intensive | transplant |
| | | | | | | chemotherapy with | intensive |
| | | | | | | HSCT | chemotherapy |
| XXXXX | XX/XX/XXXX | XX/XX/XXXX | XX | Yes | XX/XX/XXXX | XXX | XX/XX/XXXX |

### Same listing for (no listing if empty):

- Kinase
- ImiD
- ...

LYSARC 

### 6 REFERENCES

- Regression Methods in Biostatistics; Linear, Logistic, Survival, and Repeated Measures Models –
  Eric Vittinghoff, David V. Glidden, Stephen C. Shiboski, Charles E. McCulloch Statistics for Biology
  and Heath Springer
- 2. Modeling Survival Data; Extending the Cox model Terrry M. Therneau, Patricia M. Grambsch Statistics for Biology and Heath Springer
- Méthodes biostatistiques appliquées à la recherche clinique en cancérologie Andrew Kramar et Simone Mathoulin-Pélissier – L'innovation thérapeutique en cancérologie – John Libbey Eurotext

LYSARC 

### 7 APPENDICES

### 7.1 Demographic and other baseline characteristics

Table 5.12-1 Clinical examination at baseline - Included Set

| | Included Set |
|----------------------------------|--------------|
| | N=XX |
| Clinical examination at baseline | |
| Normal | XX (XX.X%) |
| Abnormal | XX (XX.X%) |
| Not done | XX (XX.X%) |
| If Abnormal, specify | |
| Due to active lymphoma | XX (XX.X%) |
| XXXXX | XX (XX.X%) |
| Due to study treatment | XX (XX.X%) |
| XXXXX | XX (XX.X%) |
| Due to other reason | XX (XX.X%) |
| XXXXX | XX (XX.X%) |

#### Listing 5.12-1 Patients with abnormal electrocardiogram at baseline – Included Set (XX patients)

| Patient identification | Inclusion date | | Electrocardiog | ram |
|---|---|---|---|---|
| number | | Date | Result | If abnormal, specify |
| XXXXX | XX/XX/XX | XX/XX/XX | Abnormal | XXXXX |

### Listing 5.12-2 Patients with other important exams performed at baseline – Included Set (XX patients)

| Patient identification number | Inclusion date | Oth | er important e | xams |
|---|---|---|---|---|
| | | Number | Description | Date |
| XXXXX | XX/XX/XX | 1 | XXXXX | XX/XX/XX |
| | | 2 | XXXXX | XX/XX/XX |

Table 5.12-2 Prior cancer history at baseline – Included Set

| | Included Set |
|--------------------------------------|--------------|
| | N=XX |
| Patients with prior cancer history | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, number of cancer per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1 ; Q3 | XX;XX |
| Min ; Max | XX ; XX |

### Listing 5.12-3 Prior cancer history at baseline – Included Set (XX patients)

| Patient | Inclusion | Prior cancer history | | | |
|---|---|---|---|---|---|
| identification | date | Number | Type of prior | Start date | End date |
| number | | | cancer | | |
| XXXXX | XX/XX/XX | XX | XXXXX | XX/XXXX | XX/XXXX |

Table 5.12-3 Relevant medical history at baseline – Included Set

| | Included Set |
|----------------------------------------|--------------|
| | N=XX |
| Patients with relevant medical history | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, number of disease per patient | |
| N | XX |
| Missing | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1;Q3 | XX;XX |
| Min ; Max | XX ; XX |

LYSARC 

Listing 5.12-4 Relevant medical history at baseline – Included Set (XX patients)

| Patient | Inclusion | Relevant medical history | | | |
|---|---|---|---|---|---|
| identification | date | Number | Type of disease | Start date | Persisting |
| number | | | | | |
| XXXXX | XX/XX/XX | XX | XXXXX | XX/XXXX | XX |

Table 5.12-4 Serology at baseline – Included Set

| 1 abic 3.12-4 Selviug | sy at basellile – ilitiaueu |
|-------------------------------|-----------------------------|
| | Included Set |
| | N=XX |
| HIV serology | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not Done | XX (XX.X%) |
| HCV serology | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not Done | XX (XX.X%) |
| HBV serology (HBs Ag) | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not Done | XX (XX.X%) |
| HBV serology (anti HBs) | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not Done | XX (XX.X%) |
| HBV serology (anti HBc) | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not Done | XX (XX.X%) |
| HBV vaccination | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| Unknown | XX (XX.X%) |
| Result of PCR for viral DNA o | f BV |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not Done | XX (XX.X%) |

Table 5.12-5 Female childbearing status - Included Set

| | Included Set<br>N=XX |
|-------------------------------------|----------------------|
| | IN-AA |
| Is female of childbearing potential | |
| No | XX (XX.X%) |
| Yes | XX (XX.X%) |
| If yes, result of pregancy test | |
| Negative | XX (XX.X%) |
| Positive | XX (XX.X%) |
| Not Done | XX (XX.X%) |

LYSARC 

## 7.2 Evaluation during study

Listing 5.12-1 Patients with abnormal clinical exam during treatment – Safety Set (XX patients)

| 0 - | | | | | | | · | |
|---|---|---|---|---|---|---|---|---|
| Patient | Inclusion | | Clinical exam | | | | | |
| identification | date | Period | Date | Result | Due to | Due to study | Due to other | Specify |
| number | | | | | Lymphoma | treatment | reason(s) | |
| XXXXX | XX/XX/XX | XX | XX/XX/XXXX | Abnormal | XX | XX | XX | XX |

## 7.3 Appendix A: Calculation of total dose and PPD

Percentage of Planned Dose is defined as follow:

$$PPD = \frac{\text{Total dose taken in mg/m}^2}{\text{Total dose expected in mg/m}^2} \times 100$$

Table 7.6-1 Calculation of total dose taken and expected

| | Total dose taken | Total dose expected |
|---|---|---|
| Cycle i | Sum of doses administered during Cycle i | Sum of doses expected during Cycle i |
| Cycle i - Cycle j | Sum of doses administered from Cycle i to Cycle j | Sum of doses expected from Cycle i to Cycle j when administered |

Table 7.6-2 Expected dose for cycle 1 according to the protocol

| Chemotherapy regimen | Dose | D1 | D2 | D3 | D4 | D8 | D15 |
|---|---|---|---|---|---|---|---|
| Dexamethasone | 40mg | Χ | Х | Х | Х | | |
| GA-101 IV | 1000mg | Χ | | | | Х | Х |
| Aracytine IV (every 12 hours) | 2 g/m <sup>2</sup> | ХХ | | | | | |
| Cisplatinum* IV | 100 mg/m <sup>2</sup> | Χ | | | | | |

Table 7.6-3 Expected dose for cycle 2 to 4 according to the protocol

| Chemotherapy regimen | Dose | D1 | D2 | D3 | D4 |
|-------------------------------|-----------------------|----|----|----|----|
| Dexamethasone | 40mg | Х | Х | Х | Х |
| GA-101 IV | 1000mg | Х | | | |
| Aracytine IV (every 12 hours) | 2 g/m <sup>2</sup> | хх | | | |
| Cisplatinum* IV | 100 mg/m <sup>2</sup> | Х | | | |

LYSARC 

# 7.4 Appendix B: MCL International Prognostic Index (MIPI) and combined biological Index (MIPIb)

Source: Hoster E et al. A new prognostic index (MIPI) for patients with advanced-stage mantle cell lymphoma. Blood 2008; 111:558-565. Erratum in: Blood 2008;111(12):5761.

MIPI Score = 0.03535 x age (years)

- + 0.6978 (if ECOG PS > 1, otherwise 0)
- + 1.367 x log<sub>10</sub>(LDH/ULN)
- + 0.9393 x log<sub>10</sub>(WBC count per 10<sup>-6</sup> L)

 $MIPI_b$  Score = 0.03535 x age (years)

- + 0.6978 (if ECOG PS > 1, otherwise 0)
- $+ 1.367 \times log_{10}(LDH/ULN)$
- + 0.9393 x log<sub>10</sub>(WBC count per 10<sup>-6</sup> L)
- + 0.02142 x Ki67 (%)

ECOG: ECOG performance status, LDH: lactate dehydrogenase, log<sub>10</sub>: logarithm with respect to base 10, ULN: upper limit of the normal range, LDH/ULN: LDH divided by ULN, WBC: white blood cell, Ki67: cell proliferation.

Risk groups are defined by:

| MIPI risk group | MIPI score | MIPI <sub>b</sub> score |
|-------------------|-----------------|-------------------------|
| Low risk | < 5.7 | < 5.7 |
| Intermediate risk | ≥ 5.7 and < 6.2 | ≥ 5.7 and < 6.5 |
| High risk | ≥ 6.2 | ≥ 6.5 |

LYSARC 

## 7.5 Appendix C: Response Criteria for Lymphoma – Lugano Classification

Bruce D. Cheson, Richard I. Fisher, Sally F. Barrington, Franco Cavalli, Lawrence H. Schwartz, Emanuele Zucca, and T. Andrew Lister. J Clin Oncol 2014;32(27):3059-68.

| Revised Criteria for Response Assessment | | |
|---|---|---|
| Response and Site | PET-CT-Based Response | CT-Based Response |
| Complete | Complete metabolic response | Complete radiologic response (all of the following) |
| Lymph nodes and extralymphatic sites | Score 1, 2, or 3_ with or without a residual mass on 5 Point Scale† It is recognized that in Waldeyer's ring or extranodal sites with high physiologic uptake or with activation within spleen or marrow (eg, with chemotherapy or myeloid colony-stimulating factors), uptake may be greater than normal mediastinum and/or liver. In this circumstance, complete metabolic response may be inferred if uptake at sites of initial involvement is no greater than surrounding normal tissue even if the tissue has high physiologic | Target nodes/nodal masses<br>must regress to ≤ 1.5 cm in LD<br>No extralymphatic sites of<br>disease |
| Nonmeasured<br>lesion<br>Organ enlargement<br>New lesions<br>Bone marrow | uptake Not applicable Not applicable None No evidence of FDG-avid disease in marrow | Not applicable Regress to normal None Normal by morphology; if indeterminate, IHC negative |

LYSARC 

| Partial | Partial metabolic response | Partial remission (all of the |
|---|---|---|
| Lymph nodes and extralymphatic sites | Score 4 or 5† with reduced uptake compared with baseline and residual mass(es) of any size At interim, these findings suggest responding disease At end of treatment, these findings indicate residual disease | following) ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites When a lesion is too small to measure on CT, assign 5 mm x 5 mm as the default value When no longer visible, 0 x 0 mm For a node > 5 mm x 5 mm, but |
| Nonmeasured<br>lesion | Not applicable | smaller than normal, use actual measurement for calculation Absent/normal, regressed, but |
| Organ enlargement New lesions | Not applicable None | no increase Spleen must have regressed by > 50% in length beyond normal |
| New lesions Bone marrow | Residual uptake higher than uptake in normal marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed). If there are persistent focal changes in the marrow in the context of a nodal response, consideration should be given to further evaluation with MRI or biopsy or an interval scan | None<br>Not Applicable |
| No Response or | No metabolic response | Stable Disease |
| Target nodes/nodal<br>masses, extranodal<br>lesions | Score 4 or 5 with no significant change in FDG uptake from baseline at interim or end of treatment | < 50% decrease from baseline<br>in SPD of up to 6 dominant,<br>measurable nodes and<br>extranodal sites; no criteria for<br>progressive disease are met |
| Nonmeasured<br>lesion | Not applicable Not applicable | No increase consistent with progressionNo increase consistent with progression |
| Organ enlargement New lesions Bone marrow | None No change from baseline | None Not applicable |
| Progressive | Progressive Metabolic Response | Progressive disease requires |
| disease Individual target | Score 4 or 5 with an increase in intensity of uptake from baseline and/or | at least 1 of the following: PPD progression |
| nodes/nodal<br>masses<br>Extranodal lesions | New FDG-avid foci consistent with lymphoma at interim or end-of-treatment assessment | An individual node/lesion must<br>be abnormal with:<br>LDi > 1.5 cm and<br>Increase by ≥ 50% from PPD |

LYSARC 

| | None | 1.0 cm for lesions > 2 cm In the setting of splenomegaly, the splenic length must increase by > 50% of the extent of its prior increase beyond baseline (eg, a 15-cm spleen must increase to > 16 cm). If no prior splenomegaly, must increase by at least 2 cm from baseline New or recurrent splenomegaly New or clear progression of preexisting nonmeasured lesions |
|---|---|---|
| Nonmeasured<br>lesion<br>New lesions | New FDG-avid foci consistent with lymphoma rather than another etiology (eg, infection, inflammation). If uncertain regarding etiology of new lesions, biopsy or interval scan may be considered New or recurrent FDG-avid foci | Regrowth of previously resolved lesions A new node > 1.5 cm in any axis A new extranodal site >1.0 cm in any axis; if < 1.0 cm in any axis, its presence must be unequivocal and must be attributable to lymphoma Assessable disease of any size unequivocally attributable to lymphoma |
| Bone Marrow | | New or recurrent involvement |

LYSARC 